CLINICAL TRIAL: NCT02587442
Title: A Phase I Study to Evaluate the Safety and Pharmacokinetics of RadProtect® in Healthy Volunteers
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of RadProtect® in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Original BioMedicals Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OBM-A01-H001
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Acute Radiation Syndrome
Keywords: Acute Radiation Syndrome; ARS; Amifostine; Radio-protectants
MeSH Terms: conditions — Acute Radiation Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RadProtect® (Experimental): RadProtect® is not a full-closed micelle, and uses ferrous iron to provide linkage between PEG-b-PGA and amifostine. Transferrin and other related proteins can chelate with ferrous iron and break the micelle releasing amifostine into the blood stream.
  Interventions: Drug: RadProtect®

INTERVENTIONS:
Drug: RadProtect® — This study will evaluate RadProtect® at sequential, escalating dose levels. Once administration is given, study subjects will be followed during 24 hours of hospitalization according to the final injection timing. All subjects will need to return to the hospital for monitoring at 7+2 days after dosing, and follow-up visits by telephone at Day 3, Day 14+2, and Day 28+2 days will need to be conducted.

SUMMARY:
This is a Phase 1, non-randomized, sequential-cohort, dose escalation, open-label study designed to evaluate the safety and tolerability of RadProtect® in healthy volunteers. This study is to be conducted at two clinical centers and in conformity with Good Clinical Practice (GCP).

ELIGIBILITY:
Inclusion Criteria:

* Each subject must be willing and able to provide written informed consent for the study
* Healthy volunteer subjects of both genders, aged 18-64 years old, and any race/ethnicity
* Subjects with normal blood pressure (between ranges of 120-140/60-80 mmHg) at screening and baseline
* Subjects with a body mass index (BMI) 18-30 kg/m2
* Men or woman of childbearing potential using adequate contraception (oral contraceptives, intrauterine device or barrier method of contraception in conjunction with spermicidal jelly, or surgically sterile) during screening, while receiving the investigational drug, and for 60 days after stopping the investigational drug
* Female subjects of childbearing potential must have a negative urine pregnancy test at screening
* Subjects with physiological examination and laboratory values within normal limits (CBC/differential, blood chemistry, iron, Total Iron Binding Capacity (TIBC), urinalysis, ECG and vital signs)
* Subjects with the ability to comprehend and complete the telephone visits, screening, and site visits
* Subjects must be able to adhere to dose and visit schedules
* Subjects who agree to abstain from taking unauthorized medications or supplements or participating in any other clinical trial or experimental treatment during this trial.

Exclusion Criteria:

* Subjects with any allergic reaction or sensitivity to glutamate acid, polyethylene glycol, or any component of the test article product
* Subjects who consume > five alcoholic beverages per week
* Subjects who are pregnant or lactating
* Subjects who have blood (or urine) levels outside the normal range for any hepatic, renal, hematologic, lipid or coagulation parameters measured.
* Subjects on Hormone Replacement Therapy within the past three months
* Subjects in any other clinical trial or experimental treatment in the past three months
* Subjects with a history of diabetes (Type 1 or Type 2 diabetes mellitus) or other endocrine disorders, hypertension, hypotension or systolic blood pressure below 80 mmHg, prior cerebrovascular accident or seizure disorder, cardiovascular, hepatic or renal disease, active cancer, hematologic disorder, thromboembolic disease, or HIV infection.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability profile including the dose limiting toxicity (DLT) of RadProtect® intravenous injection to healthy volunteers. | Day 0~ Day 28
  DLT is defined as a subject's symptom worse than a Grade 2, with the exception of the value for Total Protein and Cholesterol that should be determined by the investigator as these values may be affected by diet and there may be no discomfort or immediate risk for subjects. During the telephone visits on Day 3, 14+2, and 28+2 after injection, the study coordinator will confirm the subject's status, report to the investigators, and will schedule extra hospital visits if necessary.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters of RadProtect® by analyzing subjects' serum for free WR-1065 at different time points. | Day 0 ~ Day 1 (24 hours after dosing)
  PK samples will be obtained from the arm opposite the side of infusion. A total of approximately 4 mL of whole blood per collection time point per subject will be collected for the PK analysis. There will be a total of 10 or 16 times during this study when the sampling times for PK analysis will take place (this will depend on the dosing group).

CONTACTS AND LOCATIONS:
Locations (1):
- SNBL Clinical Pharmacology Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Chen CH, Kuo ML, Wang JL, Liao WC, Chang LC, Chan LP, Lin J. CCM-AMI, a Polyethylene Glycol Micelle with Amifostine, as an Acute Radiation Syndrome Protectant in C57BL/6 Mice. Health Phys. 2015 Sep;109(3):242-8. doi: 10.1097/HP.0000000000000326. PMID 26222219